CLINICAL TRIAL: NCT04521582
Title: Management of Hypertension Utilizing Trained Community Health Worker in Rural Municipalities of Nepal (MUTU) Study
Brief Title: Management of Hypertension Utilizing Trained Community Health Worker in Rural Municipalities of Nepal
Acronym: MUTU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Nepal Development Society (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB00011513; 744 - 2019 (Other: Nepal Health Research Council)
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Hypertension,Essential
Keywords: Hypertension; Community Health Worker; Medication; Amlodipine; Nepal
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): Participants will be first screened for their blood pressure and asked a few questions to determine eligibility. For eligible participants, FCHV will visit within ~1 week and measure blood pressure again. If found high, the participant will be referred to the nearest Health Post. At the Health Posts, if FB-CHWs confirms the diagnosis of hypertension, they will prescribe amlodipine 5 mg/d according to the study protocol and ask the patient to return in ~2 weeks. If blood pressure is controlled (<140/90 mmHg) after ~2 weeks, FB-CHWs will refill amlodipine 5 mg/d for 3 months. If not, FB-CHWs will increase the dose to 10 mg/d and follow up in ~2 weeks. If still not controlled with amlodipine 10 mg, FB-CHWs will refer the patient to the Regional Hospital in Pokhara. In addition, FCHVs will visit patients' homes 3 times (at 3-, 6-, and 9-month), provide lifestyle counseling, and follow up the adherence to hypertension treatment.
  Interventions: Drug: Amlodipine; Behavioral: Lifestyle counselling
- Comparison Group (Active Comparator): Participants will be first screened for their blood pressure and asked a few questions to determine eligibility. For eligible participants, FCHV will visit within a week or so and measure the blood pressure again. If found high, the participant will be referred to a healthcare facility ("the usual care") which can diagnose and manage hypertension. In addition, FCHVs will visit patients' homes once (around 3-month), provide lifestyle counseling, and follow up the adherence to hypertension treatment.
  Interventions: Behavioral: Lifestyle counselling

INTERVENTIONS:
Drug: Amlodipine — The facility-based community health worker will receive protocol-driven training to initiate amlodipine for hypertensive patients. These patients will receive lifestyle counseling by Female Community Health Volunteer through home visits (5 times [including baseline and end of the study] in the active municipality and 3 times [including baseline and end of the study] in the control municipality).
  Arms: Active Group
Behavioral: Lifestyle counselling — Female Community Health Volunteer will provide lifestyle counseling at the participant's home

SUMMARY:
The investigators will evaluate whether a system involving Female Community Health Volunteers (FCHVs) and facility-based community health workers (FB-CHWs) of Health Post (Auxiliary Health Workers, Auxiliary Nurse Midwives and Health Assistant) can contribute to improving hypertension care in rural Nepal. This study will be conducted in Rupa (active group) and Biruwa (comparison group) Rural Municipality of Gandaki province and enroll at least 736 hypertensive adults (322 in Rupa Rural Municipality and 414 in Biruwa Rural Municipality) who are aged 25-70 years, not taking antihypertensive medication, not pregnant and not breastfeeding, free of prior cardiovascular disease, chronic kidney disease, and diabetes. In Rupa Municipality, eligible participants will be able to receive amlodipine, one of the most frequently used antihypertensive medications, from FB-CHWs at Health Posts and five times (including baseline and end of study) of lifestyle counseling by FCHVs, whereas participants in Biruwa Municipality will receive the usual care plus three times (including baseline and end of study) of lifestyle counseling by FCHVs.

DETAILED DESCRIPTION:
Despite a large body of evidence on the effectiveness of hypertension treatment in reducing cardiovascular morbidity and mortality, the control rate of hypertension is low in many low and middle-income countries. The shortage of skilled workforce diagnosing and managing hypertension is one of the major barriers. A promising option is to involve community health workers (CHWs) in hypertension care, who have shown promising results for improving maternal and child health. However, the evidence on whether CHWs can diagnose and treat hypertension under the supervision of a physician has not been systematically tested.

Thus, this study will evaluate whether existing Facility Based-Community Health Workers (FB-CHWs) and Female Community Health Volunteers (FCHVs) of the Ministry of Health can safely and effectively diagnose hypertension and initiate/maintain protocol-based hypertension treatment. This study will be conducted in Rupa (active group) and the Biruwa (comparison group) Rural Municipality of Gandaki province. All adults aged 25-70 years of age who reside in the Rupa and Biruwa municipalities are eligible for the initial screening by data enumerators of the Nepal Development Society (NeDS). Only eligible participants who meet the inclusion criteria will participate in the study.

Rupa Rural Municipality will allow the initiation of antihypertensive medication (amlodipine) by FB-CHW at Health Posts under the supervision of a study physician. Biruwa Rural Municipality will follow usual care, which is a referral to healthcare facilities currently providing hypertension care. FCHVs will provide lifestyle counseling and follow up the adherence to hypertension treatment three times in Rupa Rural Municipality and once in Biruwa Rural Municipality.FCHV in Rupa Rural Municipality will make three home visits (at 3, 6, and 9 months) whereas FCHV in Biruwa Rural Municipality will make one home visit after 3 months of baseline. The end of the study survey will be carried out after one year by FCHV and NeDS data enumerators. The primary study outcome is a net change in systolic blood pressure among hypertensive participants 12-months after confirming hypertension in the active vs. the comparison group.

ELIGIBILITY:
Inclusion criteria

* Between 25-70 years old
* Systolic blood pressure 140-179 mmHg or diastolic blood pressure 90-119 mmHg
* Do not have a plan to leave the study municipality within a year

Exclusion criteria

* Use of antihypertensive medication in the last two weeks
* History of stroke, heart attack, heart failure, or chronic kidney disease
* History of diabetes meritus
* Pregnant or any plan to be pregnant in a year
* Breastfeeding

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1428 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Mean change in systolic blood pressure | One year
  To assess the longitudinal association of the intervention with changes in blood pressure over time, linear mixed effect models with a three-level hierarchical approach will be used.
Mean change in diastolic blood pressure | One year
  To assess the longitudinal association of the intervention with changes in blood pressure over time, linear mixed effect models with a three-level hierarchical approach will be used.

SECONDARY OUTCOMES:
Percentage of hypertension control (<140/90) among study participants | One year
  Systolic blood pressure <140 mmHg and diastolic blood pressure <90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Kunihiro Matsushita, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- Nepal (2):
  - Rupa Rural Municipality, Kāski̇̄, Gandaki
  - Biruwa Rural Municipality, Syāṅjā, Gandaki

IPD SHARING:
Plan to Share IPD: No